CLINICAL TRIAL: NCT01259271
Title: Single Center, Single Blind, Randomized, Sham Controlled Pilot Study Using Selective Nerve Stimulation (SNS) Signal for Nerve Modulation With Three Amplitudes (Supra-threshold, Sub-threshold and Sham)
Brief Title: Selective Nerve Stimulation (SNS) Pilot Study
Acronym: SNS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NM-FSB-1001
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Healthy; Pain
Keywords: human; nerve; modulation; Healthy human; sNCT; stimulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supra-threshold (Experimental): Supra-threshold is defined as the nerve stimulation amplitude at which a subject can tolerate sensory responses (like tingling, tapping in the thumb, index or middle fingers) but will not cause pain or duress to the subject. The intervention (TAMS device), is stimulating through tyco extended wear electrodes that are placed directly on top of non dominant hand healthy median nerve fibers and they feel the paresthesia or tingling sensation.
  Interventions: Device: Selective Nerve Stimulation (SNS) stimulator device
- Sub-threshold (Experimental): Sub-threshold is defined as the nerve stimulation amplitude just below the sensory perception of the subject. The intervention (TAMS device), is stimulating through tyco extended wear electrodes that are placed directly on top of non dominant hand healthy median nerve fibers. Subjects do not feel the paresthesia or tingling sensation despite there being a signal transmitted..
  Interventions: Device: Selective Nerve Stimulation (SNS) stimulator device
- Sham Control (Sham Comparator): All subjects in the sham arm will go through the same process / experimental setup as in each of the active stimulation arms; however there will be no stimulation signal during the sham stimulation (output set and SNS box locked at 0 V). As this is the Sham control, there is no intervention but rather the intevention (TAMS device) setup (Tyco electrodes, wires and stimulator) are sent with the subject as if it were on (and just like Subthreshold arm the subjects cannot feel the stimulation). Audible alerts (to signify that the box is unplugged) will be disabled throughout the duration of the study. This sham arm will be used to assess the placebo effect caused by the stimulation and hence isolate the true effect of stimulation.
  Interventions: Device: Selective Nerve Stimulation (SNS) stimulator device

INTERVENTIONS:
Device: Selective Nerve Stimulation (SNS) stimulator device — Two hours per study visit separated by a minimum of a 20 hour wash out period between stimulations.
  Other Names: Transdermal Amplitude Modulated Signal nerve stimulation device (TAMS)

SUMMARY:
The purpose of this study is to examine if a new device, the SNS (Selective Nerve Stimulator), is effective in changing the way nerves work as pain killing drugs sometimes do. During this study, the study team will place 2 adhesive patches on the inside of one of the wrists of the non-dominant hand (if the subject is right-handed the electrodes will be placed on the subject's left wrist) of the study subject. These patches will be connected by wires (leads) to a small box with a headphone jack. This is designed to provide gentle electrical stimulation through the skin. This study will look at the amount of change from normal nerve function, the sensory effects (feeling, sensations in the body), and any changes the subject has when performing the 2 hour tests. The safety of the study device will also be evaluated.

DETAILED DESCRIPTION:
Single center, single blind, randomized, crossover design, sham controlled pilot study using Selective Nerve Stimulation (SNS) signal for nerve modulation with three amplitudes (supra-threshold,sub-threshold and sham)

The primary objective of this proof of concept study is to:

• Evaluate median nerve modulation with selective nerve stimulation amplitudes (supra-threshold, sub-threshold, and sham) by means of objective quantitative sensory tests (QST) and Sensory Nerve Conduction Threshold Tests (sNCTs) in healthy subjects.

The secondary objectives to be evaluated in this study are to:

* Establish device safety profile
* Evaluate patient reported sensory descriptions and perception during modulation

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria:

* 18 years of age or older
* Ability to provide written informed consent for participation in this study
* Ability to understand and willing to comply with all study-related procedures, such as questionnaires, diaries and follow-up visits for the study duration
* Ability to not use analgesics throughout the duration of the study

Exclusion Criteria:

* Chronic peripheral pain or diagnosed neuropathy of the median nerve or the cervical spine (C6-C8) as reported by the subject
* Use of analgesics within 3 days prior to screening / baseline visit and if the subject is unable to refrain from using any analgesics throughout their study participation
* Metal implants in the forearm
* Previous nerve damage or bone injury that led to median nerve damage
* Previous surgery for carpal tunnel release in the non-dominant study hand
* Skin irritation or active infection at or near the electrode placement sites
* Allodynia involving the patch application area
* Known history of allergic reaction to the adhesive, hydrogel or any other component of the electrode or patch
* Use of an investigational drug or device within 30 days prior to study enrollment.
* Use of Cardiac pacemaker, implantable cardioverter-defibrillators (ICD's), or other electrostimulation device
* Currently untreated abuse of drugs and/or alcohol
* Psychological or medical condition that would make the study participant unadvisable
* Uncontrolled seizures (averaging > 2 seizures/month)
* Pregnant, or planning on becoming pregnant or breastfeeding during the study period
* Co-morbid condition that could limit his/her ability to participate in the study or to comply with the follow-up requirements.
* Any known inabilities to be evaluated instrumentally by quantitative sensory testing (QST) or sensory nerve conduction threshold tests (sNCTs) for a median nerve neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2011-02-01 (Actual)

PRIMARY OUTCOMES:
Modulation of Median Nerve Perception or Nerve Physiology | > 2 weeks
  The primary effectiveness endpoints are the modulation of median nerve perception or nerve physiology as measured by:
  * QST evaluated by method of levels for vibratory perception threshold (VS) in ABeta fibers and for cold sensation threshold (CS) in alpha gamma fibers and warm sensation threshold (WS) in c fibers.
  * sNCTs Current Perception Threshold (CPT) in ABeta, Alpha gamma and c fibers (CPT2k, CPT250, CPT5 respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lilienfeld, MD, Study Chair — Codman and Shurtleff
Locations (1):
- Codman & Shurtleff, Raynham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Schmidt RA, Jonas U, Oleson KA, Janknegt RA, Hassouna MM, Siegel SW, van Kerrebroeck PE. Sacral nerve stimulation for treatment of refractory urinary urge incontinence. Sacral Nerve Stimulation Study Group. J Urol. 1999 Aug;162(2):352-7. PMID 10411037
- [Background] Katz JN, Simmons BP. Clinical practice. Carpal tunnel syndrome. N Engl J Med. 2002 Jun 6;346(23):1807-12. doi: 10.1056/NEJMcp013018. No abstract available. PMID 12050342
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Verdugo RJ, Salinas RA, Castillo JL, Cea JG. Surgical versus non-surgical treatment for carpal tunnel syndrome. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD001552. doi: 10.1002/14651858.CD001552.pub2. PMID 18843618
- [Background] Eisenberg E, Backonja MM, Fillingim RB, Pud D, Hord DE, King GW, Stojanovic MP. Quantitative sensory testing for spinal cord stimulation in patients with chronic neuropathic pain. Pain Pract. 2006 Sep;6(3):161-5. doi: 10.1111/j.1533-2500.2006.00080.x. PMID 17147592
- [Background] Naeser MA, Hahn KA, Lieberman BE, Branco KF. Carpal tunnel syndrome pain treated with low-level laser and microamperes transcutaneous electric nerve stimulation: A controlled study. Arch Phys Med Rehabil. 2002 Jul;83(7):978-88. doi: 10.1053/apmr.2002.33096. PMID 12098159
- [Background] Scholten RJ, Mink van der Molen A, Uitdehaag BM, Bouter LM, de Vet HC. Surgical treatment options for carpal tunnel syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003905. doi: 10.1002/14651858.CD003905.pub3. PMID 17943805
- [Background] Huge V, Lauchart M, Forderreuther S, Kaufhold W, Valet M, Azad SC, Beyer A, Magerl W. Interaction of hyperalgesia and sensory loss in complex regional pain syndrome type I (CRPS I). PLoS One. 2008 Jul 23;3(7):e2742. doi: 10.1371/journal.pone.0002742. PMID 18648647
- [Background] Koga K, Furue H, Rashid MH, Takaki A, Katafuchi T, Yoshimura M. Selective activation of primary afferent fibers evaluated by sine-wave electrical stimulation. Mol Pain. 2005 Mar 25;1:13. doi: 10.1186/1744-8069-1-13. PMID 15813963
- [Background] Wang N, Hui-Chan C. Effects of acupoints TENS on heat pain threshold in normal subjects. Chin Med J (Engl). 2003 Dec;116(12):1864-8. PMID 14687475
- [Background] Lozano AM. Deep brain stimulation for Parkinson's disease. Parkinsonism Relat Disord. 2001 Jul;7(3):199-203. doi: 10.1016/s1353-8020(00)00057-2. PMID 11331187
- [Background] Laxton AW, Tang-Wai DF, McAndrews MP, Zumsteg D, Wennberg R, Keren R, Wherrett J, Naglie G, Hamani C, Smith GS, Lozano AM. A phase I trial of deep brain stimulation of memory circuits in Alzheimer's disease. Ann Neurol. 2010 Oct;68(4):521-34. doi: 10.1002/ana.22089. PMID 20687206
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Ben-Menachem E, Manon-Espaillat R, Ristanovic R, Wilder BJ, Stefan H, Mirza W, Tarver WB, Wernicke JF. Vagus nerve stimulation for treatment of partial seizures: 1. A controlled study of effect on seizures. First International Vagus Nerve Stimulation Study Group. Epilepsia. 1994 May-Jun;35(3):616-26. doi: 10.1111/j.1528-1157.1994.tb02482.x. PMID 8026408
- [Background] Goadsby PJ. Neurostimulation in primary headache syndromes. Expert Rev Neurother. 2007 Dec;7(12):1785-9. doi: 10.1586/14737175.7.12.1785. PMID 18052770
- [Background] Kumar K, Taylor RS, Jacques L, Eldabe S, Meglio M, Molet J, Thomson S, O'Callaghan J, Eisenberg E, Milbouw G, Buchser E, Fortini G, Richardson J, North RB. The effects of spinal cord stimulation in neuropathic pain are sustained: a 24-month follow-up of the prospective randomized controlled multicenter trial of the effectiveness of spinal cord stimulation. Neurosurgery. 2008 Oct;63(4):762-70; discussion 770. doi: 10.1227/01.NEU.0000325731.46702.D9. PMID 18981888
- [Background] Kumar K, Nath RK, Toth C. Spinal cord stimulation is effective in the management of reflex sympathetic dystrophy. Neurosurgery. 1997 Mar;40(3):503-8; discussion 508-9. doi: 10.1097/00006123-199703000-00014. PMID 9055289
- [Background] van Voskuilen AC, Oerlemans DJ, Weil EH, de Bie RA, van Kerrebroeck PE. Long term results of neuromodulation by sacral nerve stimulation for lower urinary tract symptoms: a retrospective single center study. Eur Urol. 2006 Feb;49(2):366-72. doi: 10.1016/j.eururo.2005.11.009. Epub 2006 Jan 4. PMID 16413105
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] O'Connor D, Marshall S, Massy-Westropp N. Non-surgical treatment (other than steroid injection) for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;2003(1):CD003219. doi: 10.1002/14651858.CD003219. PMID 12535461
- [Background] Alo KM, Holsheimer J. New trends in neuromodulation for the management of neuropathic pain. Neurosurgery. 2002 Apr;50(4):690-703; discussion 703-4. doi: 10.1097/00006123-200204000-00003. PMID 11904018
- [Background] Johnson MD, Burchiel KJ. Peripheral stimulation for treatment of trigeminal postherpetic neuralgia and trigeminal posttraumatic neuropathic pain: a pilot study. Neurosurgery. 2004 Jul;55(1):135-41; discussion 141-2. PMID 15214982
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Shukla G, Bhatia M, Behari M. Quantitative thermal sensory testing -- value of testing for both cold and warm sensation detection in evaluation of small fiber neuropathy. Clin Neurol Neurosurg. 2005 Oct;107(6):486-90. doi: 10.1016/j.clineuro.2004.12.016. PMID 16202822
- [Background] Franzblau A, Werner RA, Johnston E, Torrey S. Evaluation of current perception threshold testing as a screening procedure for carpal tunnel syndrome among industrial workers. J Occup Med. 1994 Sep;36(9):1015-21. PMID 7823213
- [Background] Kanai A, Suzuki A, Okamoto H. Comparison of cutaneous anesthetic effect of 8% lidocaine spray with lidocaine patch using current perception threshold test. Pain Med. 2010 Mar;11(3):472-5. doi: 10.1111/j.1526-4637.2009.00790.x. Epub 2010 Jan 22. PMID 20113414
- [Background] Yoon SH, Merrill RL, Choi JH, Kim ST. Use of botulinum toxin type A injection for neuropathic pain after trigeminal nerve injury. Pain Med. 2010 Apr;11(4):630-2. doi: 10.1111/j.1526-4637.2010.00801.x. Epub 2010 Mar 4. PMID 20210871
- [Background] Fujiuchi A, Toga T. Pharmacological effect of capsaicin on rat avoidance behaviours elicited by sine-wave electrical stimulation of different frequencies by Neurometer. J Pharm Pharmacol. 2008 Apr;60(4):467-71. doi: 10.1211/jpp.60.4.0009. PMID 18380919